CLINICAL TRIAL: NCT06687850
Title: The Effect of Animal-Assisted Therapy on Prosocial Behavior in Children With Developmental Delay or Autism Spectrum Disorder
Brief Title: Animal-Assisted Therapy in Pediatric Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Michele Kilmer, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2201382953
Record Dates: First submitted 2024-11-05; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Autism; Developmental Delay (Disorder); Behavioral Concerns
Keywords: animal-assisted therapy; canine-assisted therapy; pediatric autism spectrum disorder; verbality; prosocial behavior; emotional regulation
MeSH Terms: conditions — Developmental Disabilities; Altruism; Emotional Regulation | interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A therapy/service canine was used during therapy sessions (Experimental): The canine was included during therapy sessions and the effect of the canine on children with varying verbality was examined both during and after sessions
  Interventions: Behavioral: animal assisted therapy

INTERVENTIONS:
Behavioral: animal assisted therapy — The canine was included in therapy sessions to determine the effect of the canine on prosocial behavior and emotional regulation in autistic children with varying verbality.

SUMMARY:
The purpose of this research is to evaluate the effect of animal-assisted therapy (AAT) on prosocial behavior and emotional regulation in children with developmental delay, behavioral concerns, or autism spectrum disorder. Service dog use in the pediatric population who have these concerns is increasing and more studies are indicated to determine best practice for incorporating canines into traditional therapy sessions to enhance therapeutic outcomes. The hypothesis for this study is that inclusion of the canine will enhance therapy sessions and produce a lasting effect on prosocial behavior and emotional regulation after AAT sessions have concluded.

DETAILED DESCRIPTION:
Investigators are determining if a child's verbality affects interaction with the canine or changes the effect of animal-assisted therapy on prosocial behavior and emotional regulation in autistic children.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the program for ASD diagnostic evaluation based on their development and behavior. Could have ASD, developmental delay, or behavioral concerns.

Exclusion Criteria:

* Afraid or allergic to canines

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Targets of interaction during AAT sessions | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  * Child's caregiver: child's legal guardian or representative over age 16 years who was present during AAT sessions.
  * Therapist: Canine handler and therapist conducting the sessions.
  * Canine: Canine trained as a therapy and service dog.
  * Control objects: Defined as any inanimate object that is included in the study as a control condition for the canine
Human Interactive behaviors during AAT sessions | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Every instance of Social Communication or interactive behavior must engage a target (person, canine, or object). Interactive behaviors that occur between the primary participant and another person (caregiver or therapist) are considered Social Communication. Social Communication can be spontaneous or triggered by the initiation of another person. Interactive behaviors that occur between the primary participant and the canine or control object are considered Environmental Interactions. Subdomains include Talk, Gestures, Look, Touch, Affection, and Prosocial.
Social Communication | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Interactive behaviors that occur between the primary participant and another person (caregiver or therapist) were considered Social Communication. Social Communication could be spontaneous or triggered by the initiation of another person. Subdomains include Talk, Gestures, Look, Touch, Affection, and Prosocial.
Environmental Interactions | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Interactive behaviors that occur between the primary participant and the canine or control object are considered Environmental Interactions. Subdomains in Talk, Gestures, Look, Touch, Affection, and Prosocial.
Emotional Displays | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Emotional displays can be captured by assessing the facial expression and/or verbal content of the primary participant. Emotional display codes include Facial Emotional Display such as Smiling and Laughing, Negative Displays, No Display, or Obscured, indicating displays were not codable because they are obscured on the camera. Emotional display codes are not mutually exclusive, as many can occur within the same 10-second coding interval.
Verbal Emotional Displays | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Verbal Emotional Displays include positive, negative, or no display. This includes the content of the speech but not the tone of speech or the facial expression of the participant. If audible speech was coded under "Talk," but there are no distinguishable words, we did not code verbal emotional display. Any single statement can be coded as: (1) Positive, (2) Negative, (3) Positive and Negative, or (4) None.
Interfering Behaviors | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Interfering Behaviors coded with the OHAIRE encompass behaviors that may impair the individual's ability to participate in and benefit from an activity or interaction. These behaviors include Aggression, Overactivity, and Isolation.
Human canine interaction | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  The 3-AAT Observation ethogram was also used to code human canine interaction during AAT sessions. The revised ethogram appraises the frequency of six domains of human interaction (Affection, Play, Care, Communication, Comfort, Withdrawal) and 24 subdomains of human behavior that can occur in an AAT session. The ethogram assesses the Frequency, Intensity, and Duration of the interactions between the canine and participants.
Affection | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Affection is defined by positive behavior occurring between participants and the canine during scheduled play time incorporated into each session. Affection has two subdomains: Laughing and Petting. Intensity of Affection ranges from None (0) to Severe (4).
Laughing | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Laughing is defined as the participant laughing while playing with the canine. Audible laughter may be quiet or loud and with or without vocalization. The minimum requirement for vocalized laughter is one laugh. The minimum requirement for non-vocalized or silent laughter is two laughs with body movement such as shoulders moving to distinguish laughter from heavy breathing or sniffling.
  None (0) indicates the participant did not laugh.
  Very Mild (1) indicates the participant smiles widely showing teeth but does not audibly laugh.
  Mild (2) indicates the participant audibly once or inaudibly by moving shoulders up and down at least one time.
  Moderate (3) indicates the participant audibly two times or more or moves shoulders up and down more than twice.
  Severe (4) indicates the participant laughs more than 5 times or moves shoulders up and down more than 5 times.
Petting | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Petting is defined as the participant physically pets the canine while playing in a positive context and manner. Intensity of Petting ranges from None (0) to Severe (4).
  None (0) indicates the participant did not pet the canine during play.
  Very Mild (1) indicates the canine's skin and fur are lightly grazed when petted by participant.
  Mild (2) indicates light but clearly flush with the skin/fur of the canine. Skin and fur are lightly stretched/ shifted.
  Moderate (3) indicates more vigorous petting, fast back and forth, and skin/fur are visibly stretched/ shifted.
  Severe (4) indicates petting is very rapid, quicker back and forth, skin is very stretched, and fur is very shifted
Play | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Play is defined by the participant and canine interacting in a specific activity to promote socialization. Play has three subdomains: Fetch, Hide and Seek, and Puzzles. Intensity of Play ranges from None (0) to Severe (4).
Fetch | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Fetch is defined as the participant throwing an object, such as a ball or frisbee, in order for the canine to retrieve the object and bring the object back to the participant. This activity occurs during the scheduled play time of each session and can occur inside the clinic or outside in a grassy area in the back of the clinic. Intensity of Fetch ranges from None (0) to Severe (4).
  None (0) indicates the participant did not play fetch with the canine.
  Very Mild (1) indicates the participant played fetch for less than 10 seconds.
  Mild (2) indicates the participant played fetch for 10-30 seconds.
  Moderate (3) indicates the participant played fetch for 30-60 seconds
  Severe (4) indicates the participant played fetch for over 60 seconds
Hide and Seek | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Hide and Seek is defined as the participant playing hide and seek with the canine, either hiding themselves for the canine to find or hiding an object, such as a ball or treat, for the canine to find. This activity occurs during the scheduled play time of each session and can occur inside the clinic or outside in a grassy area in the front or back of the clinic. Intensity of Hide and Seek ranges from None (0) to Severe (4).
  None (0) indicates the participant did not play hide and seek with the canine.
  Very Mild (1) indicates the participant played hide and seek for less than 30 seconds.
  Mild (2) indicates the participant played hide and seek for 30-60 seconds.
  Moderate (3) indicates the participant played hide and seek for 60-90 seconds.
  Severe (4) indicates the participant played hide and seek for more than 90 seconds.
Puzzles | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Puzzles is defined as the participant hiding a treat in a puzzle for the canine to solve in order to get the treat. Puzzles may occur during the scheduled play time or during the scheduled seated work time during the sessions. Intensity of Puzzles ranges from None (0) to Severe (4).
  None (0) indicates the participant did not play puzzles with the canine.
  Very Mild (1) indicates the participant played puzzles for less than 30 seconds.
  Mild (2) indicates the participant played puzzles for 30-60 seconds.
  Moderate (3) indicates the participant played puzzles for 60-90 seconds.
  Severe (4) indicates the participant played puzzles for more than 90 seconds.
Care | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Care is defined as prosocial interactions initiated by participants to assist the canine. Care may occur during the scheduled play time or during the scheduled seated work time during the sessions. Care has two subdomains: Brush and Walking. Intensity of Care ranges from None (0) to Severe (4).
Brush | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Brush is defined by the participant using a brush to stroke the canine's coat. Brush may occur during the scheduled play time or during the scheduled seated work time during the sessions Intensity of Brush ranges from None (0) to Severe (4).
  None (0) indicates the participant did not brush the canine's coat.
  Very Mild (1) indicates the participant brushed the canine's coat for less than 30 seconds.
  Mild (2) indicates the participant brushed the canine's coat for 30-60 seconds.
  Moderate (3) indicates the participant brushed the canine's coat for 60-90 seconds.
  Severe (4) indicates the participant brushed the canine's coat for more than 90 seconds.
Walking | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Walking is defined as the participant walking the canine while holding the canine's leash. Walking may occur during the scheduled play time or during the scheduled seated work time during the sessions. Walking can occur inside the clinic or outside in a grassy area in the front or back of the clinic. Intensity of Walking ranges from None (0) to Severe (4).
  None (0) indicates the participant did not walk the canine using a leash.
  Very Mild (1) indicates the participant walked the canine using a leash for less than 30 seconds
  Mild (2) indicates the participant walked the canine using a leash for 30-60 seconds.
  Moderate (3) indicates the participant walked the canine using a leash for 60-90 seconds.
  Severe (4) indicates the participant walked the canine using a leash for more than 90 seconds.
Communication | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Communication is defined as words spoken by the participant directly to the canine. Communication may occur during the scheduled play time or during the scheduled seated work time during the sessions. Communication has three subdomains: Name, Command, and Verbal Affirmation. Intensity of Communication ranges from None (0) to Severe (4).
Name | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Name is defined as the participant saying the canine's name. Name must be directed toward the canine and not the caregiver or therapist. Intensity of Name ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say the canine's name.
  Very Mild (1) indicates the participant said the canine's name once.
  Mild (2) indicates the participant said the canine's name 2 - 3 times.
  Moderate (3) indicates the participant said the canine's name 4 - 5 times.
  Severe (4) indicates the participant said the canine's name more than 5 times.
Command | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Command is defined as the participant stating a command in order for the canine to do a trick or obey the participant. Command may occur during the scheduled play time or during the scheduled seated work time during the sessions. Intensity of Command ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say a command.
  Very Mild (1) indicates the participant said one command.
  Mild (2) indicates the participant said commands 2 - 3 times.
  Moderate (3) indicates the participant said commands 4 - 5 times.
  Severe (4) indicates the participant said commands more than 5 times.
Verbal Affirmation | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Verbal Affirmation is defined as the participant saying verbal affirmations directed toward the canine. Verbal Affirmation may occur during the scheduled play time or during the scheduled seated work time during the sessions. Intensity of Verbal Affirmation ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say verbal affirmations.
  Very Mild (1) indicates the participant said one verbal affirmation.
  Mild (2) indicates the participant said two verbal affirmations.
  Moderate (3) indicates the participant said verbal affirmations 3 - 5 times.
  Severe (4) indicates the participant said verbal affirmations more than 5 times.
Comfort | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Comfort is defined as prosocial behavior occurring between participants and the canine. Comfort codes behavior occurring during the scheduled seated work time of each session. Comfort has ten subdomains: Head, Face, Back, Belly, Ears, Hugs, Kiss, Treat, Floor, and Laying. Intensity of Comfort ranges from None (0) to Severe (4).
Head | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Head is defined as the participant touching the top of the canine's head during seated work time. Intensity of Head ranges from None (0) to Severe (4).
  None (0) indicates the participant did not touch the top of the canine's head while seated.
  Very Mild (1) indicates the participant touched the canine's head once while seated.
  Mild (2) indicates the participant touched the canine's head twice while seated.
  Moderate (3) indicates the participant touched the canine's head 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's head more than 5 times while seated.
Face | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Face is defined as the participant touching the canine's face during seated work time. Intensity of Face ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's face while seated.
  Very Mild (1) indicates the participant touched the canine's face once while seated.
  Mild (2) indicates the participant touched the canine's face twice while seated.
  Moderate (3) indicates the participant touched the canine's face 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's face more than 5 times while seated.
Back | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Back is defined as the participant touching the canine's back during seated work time. Intensity of Back ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's back while seated.
  Very Mild (1) indicates the participant touched the canine's back once while seated.
  Mild (2) indicates the participant touched the canine's back twice while seated.
  Moderate (3) indicates the participant touched the canine's back 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's back more than 5 times while seated.
Belly | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Belly is defined as the participant touching the canine's belly during seated work time. Intensity of Belly ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's belly while seated.
  Very Mild (1) indicates the participant touched the canine's belly once while seated.
  Mild (2) indicates the participant touched the canine's belly twice while seated.
  Moderate (3) indicates the participant touched the canine's belly 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's belly more than 5 times while seated.
Ears | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Ears is defined as the participant touching the canine's ears during seated work time. Intensity of Ears ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's ears while seated.
  Very Mild (1) indicates the participant touched the canine's ears once while seated.
  Mild (2) indicates the participant touched the canine's ears twice while seated.
  Moderate (3) indicates the participant touched the canine's ears 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's ears more than 5 times while seated.
Hugs | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Hug is defined as the participant physically hugs the canine during seated work time. Intensity of Hug ranges from None (0) to Severe (4).
  None (0) indicates the participant did not hug the canine while seated.
  Very Mild (1) indicates the participant hugged the canine once while seated.
  Mild (2) indicates the participant hugged the canine twice while seated.
  Moderate (3) indicates the participant hugged the canine 3 - 5 times while seated.
  Severe (4) indicates the participant hugged the canine more than 5 times while seated.
Kiss | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Kiss is defined as the participant kisses the canine on his head or body during seated work time. Intensity of Kiss ranges from None (0) to Severe (4).
  None (0) indicates the participant did not kiss the canine while seated.
  Very Mild (1) indicates the participant kissed the canine once while seated.
  Mild (2) indicates the participant kissed the canine twice while seated.
  Moderate (3) indicates the participant kissed the canine 3 - 5 times while seated.
  Severe (4) indicates the participant kissed the canine more than 5 times while seated.
Treat | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Treat is defined as the participant giving the canine a treat during seated work time. Intensity of Treat ranges from None (0) to Severe (4).
  None (0) indicates the participant did not give the canine a treat while seated.
  Very Mild (1) indicates the participant gave the canine a treat once while seated.
  Mild (2) indicates the participant gave the canine a treat twice while seated.
  Moderate (3) indicates the participant gave the canine a treat 3 - 5 times while seated.
  Severe (4) indicates the participant gave the canine a treat more than 5 times while seated.
Floor | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Floor is defined as the participant sitting on the floor by the canine during the seated work time. Intensity of Floor ranges from None (0) to Severe (4).
  None (0) indicates the participant did not sit on the floor by the canine while seated.
  Very Mild (1) indicates the participant sat on the floor by the canine once while seated.
  Mild (2) indicates the participant sat on the floor by the canine twice while seated.
  Moderate (3) indicates the participant sat on the floor by the canine 3 - 5 times while seated.
  Severe (4) indicates the participant sat on the floor by the canine more than 5 times while seated.
Laying | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Laying is defined as the participant physically laying their body on the canine during the seated work time. Intensity of Laying ranges from None (0) to Severe (4).
  None (0) indicates the participant did not lay their body on the canine while seated.
  Very Mild (1) indicates the participant laid their body on the canine once while seated.
  Mild (2) indicates the participant laid their body on the canine twice while seated.
  Moderate (3) indicates the participant laid their body on the canine 3 - 5 times while seated.
  Severe (4) indicates the participant laid their body on the canine more than 5 times while seated.
Withdrawal | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Withdrawal is defined as the participant moving away from interacting from the canine. Withdrawal may occur during the scheduled play time or during the scheduled seated work time during the sessions. Withdrawal has four subdomains: Moves Away, Hides, Crying, and saying "No!" to the canine. Intensity of Withdrawal ranges from None (0) to Severe (4).
Moves Away | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Moves Away is defined as the participant physically moving away from the canine to end the interaction. Intensity of Moves Away ranges from None (0) to Severe (4).
  None (0) indicates the participant did not move away from the canine.
  Very Mild (1) indicates the participant moved away from the canine once.
  Mild (2) indicates the participant moved away from the canine twice.
  Moderate (3) indicates the participant moved away from the canine 3 - 5 times.
  Severe (4) indicates the participant moved away from the canine more than 5 times.
Hides | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Hides is defined when the participant hides their face from the canine, turns their body from the canine, or hides behind an object, such as a table, to get away from the canine. Intensity of Hides ranges from None (0) to Severe (4).
  None (0) indicates the participant did not hide from the canine.
  Very Mild (1) indicates the participant hid from the canine once.
  Mild (2) indicates the participant hid from the canine twice.
  Moderate (3) indicates the participant hid from the canine 3 - 5 times.
  Severe (4) indicates the participant hid from the canine more than 5 times.
Crying | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Crying is defined as the participant crying, with or without tears, and this behavior must be directed toward the canine. Intensity of Crying ranges from None (0) to Severe (4).
  None (0) indicates the participant did not cry with the canine.
  Very Mild (1) indicates the participant cried with the canine once.
  Mild (2) indicates the participant cried with the canine twice.
  Moderate (3) indicates the participant cried with the canine 3 - 5 times.
  Severe (4) indicates the participant cried with the canine more than 5 times.
Saying "No!" | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Saying "No!" is defined as the participant verbally stating the word "No!" to the canine to end the interaction. Intensity of "No!" ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say "No!" to the canine.
  Very Mild (1) indicates the participant said "No!" to the canine once.
  Mild (2) indicates the participant said "No!" to the canine twice.
  Moderate (3) indicates the participant said "No!" to the canine 3 - 5 times.
  Severe (4) indicates the participant said "No!" to canine more than 5 times.
Frequency | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Frequency is defined by the occurrence of one of the interactions listed on the 3-AAT Observation ethogram. Interactions were measured by a tally count of each interaction.
Duration | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Duration of the interaction was assessed by rounding either up or down to the nearest 30 second mark and coded as follows.
  * 29 seconds or under was coded as 0.5
  * 30 seconds to 1 minute 29 seconds was coded as 1
  * 1:30 to 2:29 was coded as 2
  * 2:30 to 3:29 was coded as 3
  * 3:30 to 4:29 was coded as 4
  * 4:30 to 5:29 was coded as 5
  * 5:30 to 6:29 was coded as 6, and so on.
Intensity | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Intensity of the interaction was coded from None (0) to Severe (4). The mode of the interaction codes was entered to run the analysis.
Talk | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Talk is defined as verbal communication that occurs when the primary participant engages in a verbal communicative attempt with a visible target. If the target is unknown or out of frame, we coded this behavior as "No." To qualify as verbal communication, there should be audible sound clearly coming from the primary participant. We used the "three rule." If we could not determine whether the participant was talking after three viewings, we coded this behavior as "No.". If the words being spoken were intelligible, we also coded Verbal Emotional Display.
Gestures | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Gestures are defined as a form of social communication that occurs when the participant engages in a communicative attempt toward a target using physical gestures. It includes sign language and any other bodily actions that are used to communicate. The aim of the gesture should be to communicate rather than to accomplish a physical task. For example, pointing to an item on the ground is a gesture, but picking an item up off the ground is not a gesture. Talk and Gesture can be coded at the same time. When that occurred, we selected the target for BOTH codes. Gesture does not include Touch.
Look | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Look occurs when the primary participant looks in the direction of a visible target. The participant's gaze should be assessed by the angle or direction of their eyes. Look can only be coded if half of the participant's face is visible (i.e., at least one eye). Regarding canines and control objects, Look should be coded if the participant is looking at any part of the canine or object. Regarding other participants, Look can only be coded if the participant is looking at the face (or general face region) of a caregiver or therapist. If the participant looked in the direction of multiple people, canines, or objects, we coded all targets that could apply.
Touch | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Touch was coded if the primary participant comes into physical contact with a target. Touch does not include Aggression. Touch should be coded when any part of the participant's body makes contact with any part of the target. If a participant's clothing was touching another person, we also code this as Touch. Receiving any object by hand was coded as touching another person (caregiver or therapist). Similarly, receiving a control object by hand was coded as touching another person (caregiver or therapist) and the control object. In the case of giving or receiving an object by hand, we also coded this behavior as Prosocial.
Affection | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Affection was coded if the participant demonstrates physical affection or emotional warmth (i.e., verbal affection) to other humans, objects, or canines.
Prosocial | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Prosocial is defined as non-verbal behavior (i.e., physical action) that is purposefully helpful to another person, canine, or object.
Strengths and Difficulties Questionnaire | The initial SDQ is completed at the beginning of the study and the follow-up version is completed every 4 weeks and at the end of the study.
  The Strengths and Difficulties Questionnaire is a brief behavioral screening questionnaire about 2- to 17-year-olds. It exists in several versions to meet the needs of researchers, clinicians and educationalists. The SDQ ask about 25 attributes, some positive and others negative. These 25 items are divided between 5 scales: Emotional Symptoms (5 items), Conduct Problems (5 items), Hyperactivity/ Inattention (5 items), Peer Relationship Problems (5 items), Prosocial Behavior (5 items). The first four domains are added together to generate a total difficulties score. There are additional questions regarding the impact of the child's behavior concerning the chronicity, distress, social impairment, and burden to others. The initial SDQ is completed by caregivers at the beginning of the study. The follow-up SDQ is completed by caregivers every 4 weeks throughout the study and contains two additional items to evaluate the perceived effect of the intervention.
Positive and Negative Affect Scale | The PANAS is administered weekly from the start to the end of the study.
  The Positive and Negative Affect Schedule or (PANAS) is a scale that consists of different words that describe feelings and emotions. The 20-item self-report assesses positive affect (PA) and negative affect (NA). PA is associated with pleasurable engagement with the environment, whereas NA reflects a dimension of general distress summarizing a variety of negative states such as anger, guilt, or anxiety. The PANAS use a 5-point scale for caregivers to select to determine if a concept applies. The final score is derived from the sum of the ten items on both the positive and negative side. Affect states include Interested, Distressed, Excited, Upset, Strong, Guilty, Scared, Hostile, Enthusiastic, Proud, Irritable, Alert, Ashamed, Inspired, Nervous, Determined, Attentive, Jittery, Active, and Afraid.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Kilmer, DNP, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kilmer M, Hong M, Randolph D, Reichel A, Huetter S, Bowden M, Kilmer C. Animal-assisted therapy in pediatric autism spectrum disorder: A case report. Nurse Pract. 2024 Mar 1;49(3):31-39. doi: 10.1097/01.NPR.0000000000000151. PMID 38386471
- See also: Website for the university's autism program — https://accessforautism.uark.edu/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT06687850/Prot_SAP_ICF_000.pdf